CLINICAL TRIAL: NCT01729442
Title: Transrectal Prostate Cancer High-Intensity Focused Ultrasound Ablation: Assessment of Tissue Destruction With Shear-wave Ultrasound Elastography
Brief Title: Assessment of HIFU-induced Prostate Necrosis With Shear-wave Ultrasound Elastography
Acronym: IDITOP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.730
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients referred for first-line prostate HIFU ablation (Other): 10 patients
  Interventions: Other: Shear-wave ultrasound elastography (SWUE)
- Patients referred for first-line HIFU hemi-ablation (Other): 10 patients
  Interventions: Other: Shear-wave ultrasound elastography (SWUE)
- Patients referred for salvage HIFU after radiotherapy (Other): 10 patients
  Interventions: Other: Shear-wave ultrasound elastography (SWUE)

INTERVENTIONS:
Other: Shear-wave ultrasound elastography (SWUE)

SUMMARY:
Transrectal High-intensity Focused Ultrasound (HIFU) is a minimally-invasive therapy for prostate cancer that is currently assessed in two indications: as a first-line treatment (either total or focal) for patients who are not eligible for surgery and as a salvage treatment of local recurrences after radiotherapy.

It has recently been shown that Contrast-Enhanced Ultrasound (CEUS) can accurately assess the position and volume of tissue destruction at the end of prostate HIFU ablation. This can provide live feedback regarding the amount of residual non ablated tissue after HIFU treatment, which could allow immediate re-treatment in case of unsatisfactory result.

CEUS requires the injection of micro-bubbles of sulphur hexafluoride (Sonovue, Bracco, Milan, Italy) which can, at least in theory, interfere with HIFU treatment. Therefore, it is necessary to wait 20 to 30 minutes before re-treating the patient.

Shear-wave ultrasound elastography (SWUE, Supersonic Imagine, Aix-en-Provence, France) can quantify tissue stiffness. Moreover, post-HIFU necrosis is known to be stiffer than undestroyed prostate tissue. Therefore, SWUE could be an alternative to CEUS, and the purpose of this study is to evaluate the accuracy of SWUE in depicting the position and volume of therapeutic necrosis after prostate cancer High-Intensity Focused Ultrasound (HIFU) ablation.

The present study is an exploratory, monocentric, prospective, descriptive study. Three groups of 10 patients with prostate cancer will be evaluated: patients referred for first-line prostate HIFU ablation, patients referred for first-line HIFU hemi-ablation (focal treatment) and patients referred for salvage HIFU after radiotherapy.

SWUE will be obtained the day before HIFU ablation (D-1), immediately after HIFU ablation (D0) and the following day (D+1). CEUS will be performed immediately after HIFU ablation and D0 SWUE.

The primary endpoint is the comparison of the thickness of undestroyed parenchyma measured by SWUE and CEUS.

The secondary endpoints are:

* The evolution of shear elasticity within the treated area measured by SWUE at D-1, D0 and D+1,
* Adverse events related to SWUE.

The study will last 40 months.

ELIGIBILITY:
Inclusion Criteria :

* Age > 18 years
* Prostate cancer proved by biopsy
* Prostate cancer not eligible for surgery referred for total or hemi HIFU ablation, OR prostate cancer local recurrence referred for salvage HIFU ablation
* Anal and rectal normal anatomy
* Life expectancy ≥ 5 years
* Satisfactory general condition (ASA 1 to 3)
* Informed consent signed
* Affiliation to the French social security system or equivalent social security system.

Exclusion Criteria:

* Patient treated by hormonotherapy
* Prostatic calcifications preventing HIFU ablation
* Distance between rectal mucosa and prostatic capsule ≥ 6 mm
* History of inflammatory bowel disease
* Sclerosis of the bladder neck or urethral stenosis
* Rectal fistula
* Ongoing urinary infection
* Impaired renal function (MDRD < 30mL/min/1,73 m²)
* Severe BPCO
* Acute endocarditis/ Hypercoagulation/ recent thromboembolism
* Latex or sulphur hexafluoride allergy
* Contraindication to the injection of Sonovue®
* Patient on protection of the Court, under supervision or trusteeship
* Inability to express an informed consent
* Patient already enrolled in a study that could interfere with this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the thickness of undestroyed parenchyma | Day 0
  Briefly, the thickness of undestroyed parenchyma will be measured on CEUS and D0 SWUE in the anterior, lateral and posterior parts of both prostatic lobes. The thickness (height) of undestroyed parenchyma left at both apex will also be measured.
  Measurements obtained with CEUS (used as reference) and SWUE will be compared.

SECONDARY OUTCOMES:
Evolution of shear elasticity in the treated area | D-1 / D0 / D+1
  Using CEUS images as reference, a Region-of-Interest (ROI) will be placed within the area destroyed by HIFU in both lobes (except for the hemi-HIFU group). The stiffness within the ROI will be measured before HIFU ablation (D-1), immediately after (D0) and the day after (D+1).
  One or two ROI will also be placed in undestroyed tissue (as shown by CEUS used as reference) and the evolution of stiffness from D-1 to D+1 will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rouvière, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France